CLINICAL TRIAL: NCT01108809
Title: Evaluation of the Effect of Telmisartan (Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg) on Blood Pressure and Cardiovascular Risk Factor Index in High Risk Hypertensive Patients
Brief Title: Evaluation of the Effect of Telmisartan on Blood Pressure Control of High Risk Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.592
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with arterial hypertension
  Interventions: Drug: Telmisartan or Telmisartan and Hydrochlorthiazide

INTERVENTIONS:
Drug: Telmisartan or Telmisartan and Hydrochlorthiazide — Telmisartan 80mg +/- Hydrochlorthiazide 12.5mg or 25mg

SUMMARY:
The study is designed to evaluate the effect of treatment with Micardis/MicardisPlus on blood pressure and its ability to reduce different indicated cardiovascular risk scores. The study will also evaluate the current antihypertensive treatment pattern in the daily practice among the patient population at increased cardiovascular risk.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of essential arterial hypertension (BP>140/90 mm HG or BP>130/80 mm Hg for diabetic patients)
* at least one additional cardiovascular risk factor and/or known single or multiple end organ damage and/or previous cardiovascular disease

Exclusion criteria:

* hypersensitivity to the active substance or to any of the excipients in any ACE inhibitor or angiotensin receptor blocker (ARB) available on the local market, as prescribed in the SPC
* pregnancy and lactation
* diseases involving biliary obstruction
* severe liver impairment
* severe hypertension
* malignant hypertension
* secondary hypertension
* patients age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with arterial hypertension
Sampling Method: Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (49):
- Romania (49):
  - Boehringer Ingelheim Investigational Site 1, Arad
  - Boehringer Ingelheim Investigational Site 5, Bacau
  - Boehringer Ingelheim Investigational Site 6, Baia Mare
  - Boehringer Ingelheim Investigational Site 9, Brasov
  - Boehringer Ingelheim Investigational Site 8, Brăila
  - Boehringer Ingelheim Investigational Site 10, Bucharest
  - Boehringer Ingelheim Investigational Site 11, Bucharest
  - Boehringer Ingelheim Investigational Site 12, Bucharest
  - Boehringer Ingelheim Investigational Site 13, Bucharest
  - Boehringer Ingelheim Investigational Site 14, Bucharest
  - Boehringer Ingelheim Investigational Site 15, Bucharest
  - Boehringer Ingelheim Investigational Site 16, Bucharest
  - Boehringer Ingelheim Investigational Site 17, Bucharest
  - Boehringer Ingelheim Investigational Site 18, Bucharest
  - Boehringer Ingelheim Investigational Site 19, Bucharest
  - Boehringer Ingelheim Investigational Site 20, Bucharest
  - Boehringer Ingelheim Investigational Site 21, Bucharest
  - Boehringer Ingelheim Investigational Site 22, Bucharest
  - Boehringer Ingelheim Investigational Site 23, Buzău
  - Boehringer Ingelheim Investigational Site 4, Campulung Muscel
  - Boehringer Ingelheim Investigational Site 42, Carei
  - Boehringer Ingelheim Investigational Site 24, Călăraşi
  - Boehringer Ingelheim Investigational Site 26, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 27, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 28, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 29, Constanța
  - Boehringer Ingelheim Investigational Site 31, Craiova
  - Boehringer Ingelheim Investigational Site 2, Curtea de Argeş
  - Boehringer Ingelheim Investigational Site 38, Drobeta-Turnu Severin
  - Boehringer Ingelheim Investigational Site 32, Galati
  - Boehringer Ingelheim Investigational Site 34, Iași
  - Boehringer Ingelheim Investigational Site 35, Iași
  - Boehringer Ingelheim Investigational Site 36, Iași
  - Boehringer Ingelheim Investigational Site 37, Iași
  - Boehringer Ingelheim Investigational Site 7, Oradea
  - Boehringer Ingelheim Investigational Site 3, Piteşti
  - Boehringer Ingelheim Investigational Site 40, Ploieşti
  - Boehringer Ingelheim Investigational Site 41, Ploieşti
  - Boehringer Ingelheim Investigational Site 49, Râmnicu Vâlcea
  - Boehringer Ingelheim Investigational Site 25, Reşiţa
  - Boehringer Ingelheim Investigational Site 33, Slobozia
  - Boehringer Ingelheim Investigational Site 43, Suceava
  - Boehringer Ingelheim Investigational Site 30, Târgovişte
  - Boehringer Ingelheim Investigational Site 39, Târgu Mureş
  - Boehringer Ingelheim Investigational Site 44, Timișoara
  - Boehringer Ingelheim Investigational Site 45, Timișoara
  - Boehringer Ingelheim Investigational Site 46, Timișoara
  - Boehringer Ingelheim Investigational Site 47, Timișoara
  - Boehringer Ingelheim Investigational Site 48, Tulcea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Started | 295
Completed | 291
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 295
Age, Continuous [Mean (Standard Deviation); unit: years] — Data on age available for 294 patients
  years | 61.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 123
Systolic Blood Pressure (mean) [Mean (Standard Deviation); unit: mmHg] | 171 (16.2)
Diastolic Blood Pressure (mean) [Mean (Standard Deviation); unit: mmHg] | 97 (10.4)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] — Data on heart rate available for 281 patients
  beats/minute | 79 (11.5)
Additional antihypertensive treatment at baseline [Number; unit: Percentage of participants] — Participants may have taken more than one antihypertensive treatment, so the percentages will not add to 100 percent.
  Percentage of participants
    ACE inhibitors | 53.1
    Diuretics | 58.6
    Calcium Channel Blockers | 35.1
    Beta Blockers | 61.9
    Other | 15.5

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline to Study End
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 292
mmHg | -39.2 (6.6)

2. Primary Outcome: Change in Diastolic Blood Pressure From Baseline to Study End
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 292
mmHg | -17.8 (2.8)

3. Primary Outcome: Evolution of the Cardiovascular Risk Factor SCORE From Baseline to Study End
Description: A 10 year risk of fatal cardiovascular disease (CVD) in populations at high risk. Minimum 0 percent risk to Maximum 47 percent risk. Investigator judgement of evolution of SCORE from baseline to end of study. (Positive = reduction in CV risk; Neutral = no change in CV risk; Negative = deterioration in CV risk; Missing = no data available)
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 295
Percentage of participants
  Positive | 64.8
  Neutral | 8.8
  Negative | 0.3
  Missing | 26.1

4. Primary Outcome: Evolution of the Cardiovascular Risk Factor Framingham From Baseline to Study End
Description: 10-year risk for hard coronary heart disease (CHD) outcomes (Myocardial Infarction and coronary death), according to Framingham Heart Study, measured in percent. Low risk (10 or less CHD risk at 10 years), intermediate risk (10-20), high risk (20 or more). Investigator judgement of evolution of Framingham risk score from baseline to end of study. (Positive = reduction in CV risk; Neutral = no change in CV risk; Negative = deterioration in CV risk; Missing = no data available)
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 295
Percentage of participants
  Positive | 58.3
  Neutral | 10.2
  Negative | 0.3
  Missing | 31.2

5. Primary Outcome: Evolution of the European Society of Hypertension / European Society of Cardiology (ESH/ESC) Based Cardiovascular Risk Factor From Baseline to Study End
Description: ESH is the European society of hypertension, and ESC is the European society of cardiology. Investigator judgement of evolution of CV risk based on ESH/ ESC criteria from baseline to end of study. (Positive = reduction in CV risk; Neutral = no change in CV risk; Negative = deterioration in CV risk; Missing = no data available)
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 295
Percentage of participants
  Positive | 65.1
  Neutral | 12.9
  Negative | 0.3
  Missing | 21.7

6. Secondary Outcome: Percentage of Patients That Achieve Target Blood Pressure Values According to the European Society of Hypertension/European Society of Cardiology (ESH/ESC)
Description: ESH/ESC a goal of treatment to be below values 130/80 mm/Hg for diabetic patients and below 140/90 mmHg for non-diabetic patients
Time Frame: Visit 3 (6 months from baseline)
Population: Patients with data at 3rd visit
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 295
Percentage of participants | 57.3

7. Secondary Outcome: Additional Antihypertensive Treatment Pattern at Visit 3 (End of Study)
Time Frame: 6 Months
Population: Patients with data at 3rd visit
Measure: Number; unit: Percentage of participants
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 201
Percentage of participants
  ACE inhibitors | 16.9
  Diuretics | 34.8
  Calcium Channel Blockers | 39.3
  Beta Blockers | 75.1
  Other | 20.9

8. Secondary Outcome: Change in Heart Rate From Baseline to Study End
Time Frame: From baseline to visit 3 (6 months)
Population: Patients with data both at baseline and on 3rd visit
Measure: Mean (Standard Deviation); unit: beats / minute
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Number analyzed (Participants) | 269
beats / minute | -7.6 (3.9)

9. Secondary Outcome: Number of Participants Not Completing Study
Description: Number of participants discontinuing study early for given reason
Time Frame: 3rd visit (6 months)
Population: Patients with data at 3rd visit
Measure: Number; unit: Number of participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 295
Number of participants
  Adverse Event | 3
  Lost to follow up | 1

10. Secondary Outcome: Number of Patients With Adverse Events (AE)
Time Frame: 6 months
Population: Treated patients
Measure: Number; unit: Number of participants
Arm/Group | Micardis® 80mg MicardisPlus® 80/12.5 mg
Number analyzed (Participants) | 295
Number of participants | 4

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg
Serious Adverse Events (participants affected / at risk) | 1/295
Other Adverse Events (participants affected / at risk) | 0/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micardis® 80 mg/ MicardisPlus® 80/12.5 mg; 80/25 mg (N=295)
Generalized angioedema (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes